CLINICAL TRIAL: NCT02314728
Title: Cervical Ripening in Premature Rupture of Membranes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Montefiore Medical Center (Other)
Responsible Party: Principal Investigator, Peter S. Bernstein, Professor, Montefiore Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2014-3462
Record Dates: First submitted 2014-12-08; First posted 2014-12-11 (Estimated); Results first posted 2021-08-10 (Actual); Last update posted 2021-08-10 (Actual); Status verified 2021-08

CONDITIONS: Pregnancy; Premature Rupture of Membranes; Preterm Premature Rupture of Membranes; Unfavorable Cervix
Keywords: Bishop Score; Induction of Labor; Cervical Ripening; Unfavorable Cervix; Mode of Delivery; C-Section; Cesarean Section; Misoprostol; Prostaglandin; Prostaglandin E1
MeSH Terms: conditions — Fetal Membranes, Premature Rupture; Preterm Premature Rupture of the Membranes | interventions — Misoprostol; Oxytocin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Misoprostol (Active Comparator): Those randomized to the prostaglandin arm will receive PGE1 (misoprostol) in a dose of 25mcg placed vaginally every 4 hours as per hospital protocol.
  Interventions: Drug: Misoprostol
- Oxytocin Alone (Active Comparator): Those randomized to the oxytocin arm will receive infusion of oxytocin, which will then be titrated per hospital protocol or until adequate contractions.
  Interventions: Drug: Oxytocin

INTERVENTIONS:
Drug: Misoprostol — Patients who are randomized to receive misoprostol will have 25mcg placed vaginally. Repeated dosing of misoprostol is based on clinical exam and clinical judgment of the provider.
  Other Names: Cytotec
  Arms: Misoprostol
Drug: Oxytocin — Patients who are randomized to receive oxytocin alone will receive intravenous administration of oxytocin as designated by the hospital protocol. Protocol begins with 2 milliunits of oxytocin that is then titrated over time. Titration is based on clinical exam and clinical judgment of the provider and is continued until there are adequate uterine contractions.
  Other Names: Pitocin
  Arms: Oxytocin Alone

SUMMARY:
Premature rupture of membranes (PROM) is diagnosed by demonstrating amniotic fluid in the vaginal canal before the onset of labor. The integrity of the amniotic membrane is compromised thereby increasing the risk of intrauterine infection and compression of the umbilical cord. PROM complicates 3% to 8% of pregnancies in the US and is responsible for 30% of preterm births. Intrauterine infection remains the most significant maternal and neonatal sequelae associated with PROM and this risk increases with the length of time from ruptured membrane to delivery. Induction of labor has been shown to reduce the rates of chorioamnionitis, endometritis and NICU admissions4. Specifically, induction of labor with prostaglandin agents followed by oxytocin, versus oxytocin alone has been shown to be effective for labor induction resulting in vaginal delivery. Management strategies for PROM have been controversial, and published studies on outcomes are over one to two decades old, which does not account for changes in clinical trends and practice patterns. Recently ACOG recommends that patients presenting at 37 weeks gestation or greater with PROM should be induced if not in labor, and "generally with oxytocin". In women with PROM without the onset of labor, the cervix is commonly unfavorable and induction with oxytocin alone may lead to an increased risk of cesarean section. With a c-section rate as high as 33%, women undergoing induction of labor have an increased risk of c-section and its associated morbidity and long term sequela. ACOG's recommendation for the use of oxytocin as the induction agent may be meant to avoid a theoretical increased risk of chorioamnionitis in this patient population however it does not take into account the status of the cervix, which may result in a increased risk of c-section. The purpose of the proposed study is to determine whether cervical ripening in women with PROM and an unfavorable cervix is associated with increase rates of vaginal delivery and decreased cesarean section rate compared to induction of labor with oxytocin alone. The investigators aim to determine the incidence of endometritis, and neonatal infection associated with PROM in the current medical environment of antibiotic prophylaxis and antenatal steroid use, taking into account the changes in patient characteristics.

DETAILED DESCRIPTION:
We will perform a prospective randomized control trial involving women with singleton gestation at ≥ 34 weeks gestation who require an induction of labor after diagnosis of PROM with an unfavorable cervix. PROM will be diagnosed and confirmed with sterile speculum examination demonstrating pooling and/or positive ferning or nitrazine. Cervical status will be assessed by visual exam, digital exam or transvaginal ultrasound to assign a Bishop score (dilation, effacement, station, consistency & position). Determination of patient eligibility will be based on the clinical exam and confirmation of PROM. Upon diagnosis, if the patient meets inclusion criteria and accepts to participate in the study, they will be consented by the study investigator and then be randomized to prostaglandin followed by oxytocin or oxytocin alone group. Allocation concealment will be performed via the utilization of pre-sequentially numbered, manila sealed envelopes stapled closed.

There are two treatment groups and will be analyzed on an intent-to-treat basis. Randomization will be performed using a computer generated simple randomization sequence. Data safety monitoring will be instituted (see data safety monitoring plan below). Once randomization is completed, the labor and delivery providers will be informed of the treatment arm and this will be placed on the chart. Those randomized to the prostaglandin arm will receive PGE1 (misoprostol) in a dose of 25mcg placed vaginally every 4 hours as per hospital protocol. Those randomized to the oxytocin arm will receive infusion of oxytocin, which will then be titrated per hospital protocol until adequate contractions. Further management after the start of the respective arm will be based on clinical judgment of the provider.

ELIGIBILITY:
Inclusion Criteria:

1. All pregnant women diagnosed with PROM without evidence of labor requiring induction
2. Gestational Age > 34 weeks
3. Bishop score < 6
4. Category I Fetal heart rate tracing

Exclusion Criteria:

1. Contraindication to Induction of Labor
2. Multiple gestation
3. Fetal Anomalies
4. Previous C-Section
5. HIV Positive Patients

Ages: 15 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 230 (Actual)
Dates: Start 2014-10-01 (Actual); Primary Completion 2016-05-30 (Actual); Study Completion 2016-05-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kafui Demasio, MD, MPH, Principal Investigator — Montefiore Medical Center
Locations (1):
- Montefiore Medical Center, The Bronx, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Merrill DC, Zlatnik FJ. Randomized, double-masked comparison of oxytocin dosage in induction and augmentation of labor. Obstet Gynecol. 1999 Sep;94(3):455-63. doi: 10.1016/s0029-7844(99)00338-5. PMID 10472877
- [Result] Dare MR, Middleton P, Crowther CA, Flenady VJ, Varatharaju B. Planned early birth versus expectant management (waiting) for prelabour rupture of membranes at term (37 weeks or more). Cochrane Database Syst Rev. 2006 Jan 25;(1):CD005302. doi: 10.1002/14651858.CD005302.pub2. PMID 16437525
- [Result] Mercer BM. Preterm premature rupture of the membranes: current approaches to evaluation and management. Obstet Gynecol Clin North Am. 2005 Sep;32(3):411-28. doi: 10.1016/j.ogc.2005.03.003. PMID 16125041
- [Result] Kunze M, Hart JE, Lynch AM, Gibbs RS. Intrapartum management of premature rupture of membranes: effect on cesarean delivery rate. Obstet Gynecol. 2011 Dec;118(6):1247-1254. doi: 10.1097/AOG.0b013e3182351b0c. PMID 22105253
- [Result] Hannah ME, Ohlsson A, Farine D, Hewson SA, Hodnett ED, Myhr TL, Wang EE, Weston JA, Willan AR. Induction of labor compared with expectant management for prelabor rupture of the membranes at term. TERMPROM Study Group. N Engl J Med. 1996 Apr 18;334(16):1005-10. doi: 10.1056/NEJM199604183341601. PMID 8598837
- [Result] Balci O, Mahmoud AS, Acar A, Colakoglu MC. Comparison of induction of labor with vaginal misoprostol plus oxytocin versus oxytocin alone in term primigravidae. J Matern Fetal Neonatal Med. 2011 Sep;24(9):1084-7. doi: 10.3109/14767058.2010.531798. Epub 2010 Nov 19. PMID 21087166
- [Result] Gonen R, Samberg I, Degani S. Intracervical prostaglandin E2 for induction of labor in patients with premature rupture of membranes and an unripe cervix. Am J Perinatol. 1994 Nov;11(6):436-8. doi: 10.1055/s-2007-994615. PMID 7857439
- [Result] Mahmood TA, Dick MJ, Smith NC, Templeton AA. Role of prostaglandin in the management of prelabour rupture of the membranes at term. Br J Obstet Gynaecol. 1992 Feb;99(2):112-7. doi: 10.1111/j.1471-0528.1992.tb14466.x. PMID 1554660
- [Result] Duff P, Huff RW, Gibbs RS. Management of premature rupture of membranes and unfavorable cervix in term pregnancy. Obstet Gynecol. 1984 May;63(5):697-702. PMID 6717874
- [Result] Vrouenraets FP, Roumen FJ, Dehing CJ, van den Akker ES, Aarts MJ, Scheve EJ. Bishop score and risk of cesarean delivery after induction of labor in nulliparous women. Obstet Gynecol. 2005 Apr;105(4):690-7. doi: 10.1097/01.AOG.0000152338.76759.38. PMID 15802392
- [Result] Wing DA, Paul RH. Induction of labor with misoprostol for premature rupture of membranes beyond thirty-six weeks' gestation. Am J Obstet Gynecol. 1998 Jul;179(1):94-9. doi: 10.1016/s0002-9378(98)70256-x. PMID 9704771
- [Result] Kenyon S, Boulvain M, Neilson JP. Antibiotics for preterm rupture of membranes. Cochrane Database Syst Rev. 2013 Dec 2;2013(12):CD001058. doi: 10.1002/14651858.CD001058.pub3. PMID 24297389
- See also: ACOG Practice Bulletin 139: Premature Rupture of Membranes — https://www.scribd.com/doc/211885423/Practice-Bulletins-No-139-Premature-Rupture-of-Membranes
- See also: ACOG Practice Bulletin 107: Induction of Labor — https://www.mnhospitals.org/Portals/0/Documents/patientsafety/Perinatal/acog--practice_bulletin_107_2009.pdf

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Women with PROM, Bishop Score <6, singleton, >/=34 weeks of gestation
Pre-assignment Details: Calculated Sample size of 208-104 per each arm. Recruited 230 women out of 294 admitted with PROM and assessed for eligibility.
Groups:
- Vaginal Misoprostol: PROM >/= 34 weeks
  Those randomized to the prostaglandin arm will receive PGE1 (misoprostol) in a dose of 25mcg placed vaginally every 4 hours as per hospital protocol.
  Misoprostol: Patients who are randomized to receive misoprostol will have 25mcg placed vaginally.
- Oxytocin Alone: PROM >/= 34 weeks
  Those randomized to the oxytocin arm will receive infusion of oxytocin, which will then be titrated per hospital protocol or until adequate contractions.
  Oxytocin: Patients who are randomized to receive oxytocin alone will receive intravenous administration of oxytocin as designated by the hospital protocol. Protocol begins with 2 milliunits of oxytocin that is then titrated over time. Titration is based on hospital protocol, clinical exam and clinical judgment of the provider and is continued until there are adequate uterine contractions to delivery.
Period: Overall Study
Arm/Group | Vaginal Misoprostol | Oxytocin Alone
Started | 117 | 113
Completed | 116 | 112
Not Completed | 1 | 1
Not completed — Protocol Violation | 1 | 0
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Vaginal Misoprostol: PROM greater than or equal to 34 weeks of gestation with unfavorable cervical examination (Bishop score </= 6.
  Women with PROM randomized to the prostaglandin arm will receive PGE1 (misoprostol) in a dose of 25 mcg transvaginal every 4 hours as per hospital protocol.
  Misoprostol: Women with PROM who are randomized to receive misoprostol will have 25 mcg placed vaginally.
- Oxytocin Alone: PROM greater than or equal to 34 weeks of gestation with unfavorable cervical examination (Bishop score </= 6.
  Women randomized to the oxytocin arm will receive infusion of oxytocin that is titrated as per hospital protocol, and until adequate uterine contractions are achieved.
  Oxytocin: Women with PROM who are randomized to receive oxytocin alone will receive intravenous administration of oxytocin as designated by the hospital protocol. The hospital protocol begins with 2 milliunits of oxytocin that is then titrated upward by 2 millunits every 20-30 minutes until adequate contractions that cause cervical change is obtained. Titration is based on hospital protocol, clinical examination and clinical judgment of the provider, and is continued until there are adequate uterine contractions that cause the cervix to change until delivery.
- Total: Total of all reporting groups
Arm/Group | Vaginal Misoprostol | Oxytocin Alone | Total
Number analyzed (Participants) | 116 | 112 | 228
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 2 | 6 | 8
  Between 18 and 65 years | 114 | 106 | 220
  >=65 years | 0 | 0 | 0
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 25.5 [18 to 43] | 26 [16 to 45] | 26.0 [16 to 45]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 116 | 112 | 228
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 10 | 9 | 19
  African American | 28 | 26 | 54
  Hispanic | 64 | 62 | 126
  Other | 14 | 15 | 29
Region of Enrollment [Number; unit: participants]
  United States | 116 | 112 | 228

OUTCOME MEASURES:

1. Primary Outcome: Rate of Cesarean Section
Description: Mode of delivery via cesarean section or vaginal delivery
Time Frame: within 48 hours
Measure: Number; unit: participants
Groups:
- Vaginal Misoprostol: PROM greater than or equal to 34 weeks of gestation
  Those randomized to the prostaglandin arm will receive PGE1 (misoprostol) in a dose of 25mcg placed vaginally every 4 hours as per hospital protocol.
  Misoprostol: Patients who are randomized to receive misoprostol will have 25mcg placed vaginally.
- Oxytocin Alone: PROM greater than or equal to 34 weeks of gestation
  Those randomized to the oxytocin arm will receive infusion of oxytocin, which will then be titrated per hospital protocol or until adequate contractions.
  Oxytocin: Patients who are randomized to receive oxytocin alone will receive intravenous administration of oxytocin as designated by the hospital protocol. Protocol begins with 2 milliunits of oxytocin that is then titrated over time. Titration is based on hospital protocol, clinical exam and clinical judgment of the provider and is continued until there are adequate uterine contractions to delivery.
Arm/Group | Vaginal Misoprostol | Oxytocin Alone
Number analyzed (Participants) | 116 | 112
participants
  Cesarean Delivery | 27 | 26
  Vaginal Delivery | 89 | 86
Statistical Analysis 1: Comparison: Vaginal Misoprostol vs Oxytocin Alone; Test type: Superiority; p = 0.99, Fisher Exact

2. Secondary Outcome: Maternal and Neonatal Infectious Morbidity
Description: Maternal infection defined as fever >100.4 on at least two occasions during labor, continued antibiotic treatment on or after PPD#1, histologic confirmation of chorioamnionitis. Dose of Oxytocin, Tachysystole, Estimated blood loss at delivery, maternal length of stay, Epidural use, Indication for cesarean delivery
  Neonatal infection defined as WBC <5000 and absolute neutrophil count <1000 or positive blood cultures and neonatal fever, NICU admission, Apgar score less than 7 at 5 minutes,
Time Frame: within 72 hours
Population: Women induced for PROM at greater than, or equal to 34 weeks of gestation with unfavorable cervical examination (Bishop score </= 6 and their neonates.
Measure: Count of Participants; unit: Participants
Arm/Group | Vaginal Misoprostol | Oxytocin Alone
Number analyzed (Participants) | 116 | 112
Participants
  NICU Admission | 13 | 15
  Histologic Chorioamnionitis: number analyzed (Participants) | 27 | 26
  Histologic Chorioamnionitis | 9 | 13
Statistical Analysis 1: Comparison: Vaginal Misoprostol vs Oxytocin Alone; NICU admission; Test type: Superiority; p = 0.60, Fisher Exact
Statistical Analysis 2: Comparison: Vaginal Misoprostol vs Oxytocin Alone; histologic chorioamnionitis; Test type: Superiority; p = 0.13, Fisher Exact

ADVERSE EVENTS:
Time Frame: 1 month
Description: In the event of adverse event a report is generated and reviewed by the monitoring committee who were the Director of Labor and Delivery and Vice Chair of Obstetrics.
Arm/Group | Misoprostol | Oxytocin Alone
All-Cause Mortality (participants affected / at risk) | 0/117 | 0/113
Serious Adverse Events (participants affected / at risk) | 0/117 | 0/113
Other Adverse Events (participants affected / at risk) | 0/117 | 0/113

LIMITATIONS AND CAVEATS:
1. Protocol breech
2. Variability in provider practices on labor and delivery. Reluctance to use misoprostol with rupture membranes.
3. Patient wait times impacted compliance with protocol. They went into labor while awaiting for a labor bed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No